CLINICAL TRIAL: NCT04435691
Title: An Open-Label Phase IB/II Study of Magrolimab in Combination With Azacitidine and Venetoclax for the Treatment of Patients With Acute Myeloid Leukemia (AML)
Brief Title: Magrolimab, Azacitidine, and Venetoclax for the Treatment of Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: 75% > Participants
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0027; NCI-2020-04163 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0027 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; magrolimab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine, venetoclax, magrolimab) (Experimental): Patients receive azacitidine SC or IV over 30-60 minutes on days 1-7, venetoclax PO QD on days 1-28 of cycle 1 (may be reduced to days 1-21 for subsequent cycles after principal investigator approval), and magrolimab IV over 2-3 hours on days 1, 4, 8, 11, 15, and 22 of cycle 1, days 1, 8, 15, and 22 of cycle 2, and days 1 and 15 of cycle 3 and subsequent cycles. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Biological: Magrolimab; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Biological: Magrolimab — Given IV
  Other Names: Hu5F9-G4
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of magrolimab and venetoclax when given together with azacitidine and to see how well they work in treating patients with acute myeloid leukemia. Magrolimab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving magrolimab, azacitidine, and venetoclax may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and maximum tolerable dose (MTD) of this combination in patients with acute myeloid leukemia (AML).

II. To determine the response rate (RR) including CR (complete remission) + CRi (complete remission with incomplete count recovery) within 3 months of treatment initiation of this combination in patients with AML.

SECONDARY OBJECTIVES:

I. To assess the CR + complete remission with partial hematological recovery (CRh) rate and morphologic leukemia free (MLF) rate within 3 months of treatment initiation of this combination in patients with AML.

II. To determine the duration of response (DOR), event-free survival (EFS), overall survival (OS), MRD status at response and best MRD response attained by flow-cytometry, 4- and 8-week mortality, and number of patients bridged to hematopoetic stem cell transplant (HSCT) and median duration to HSCT from the initiation of the combination.

III. To investigate correlations of response to this combination with a pre- therapy, on-therapy, and progression 81-gene panel of gene mutations in AML.

EXPLORATORY OBJECTIVES:

I. To investigate possible relationships between response and non-response to the combination with pretherapy, on-therapy, and progression gene expression signatures.

II. To investigate the characterization of genetic heterogeneity in tumor cell populations, by performing targeted single-cell sequencing on longitudinally collected AML tumor populations from patients using a novel microfluidic approach that barcodes amplified genomic deoxyribonucleic acid (DNA) from thousands of individual leukemia cells confined to droplets (single cell sequencing).

III. To identify individual cell populations (AML blasts, T-cells - both bulk and T-cell subsets and coreceptor/ligand expression, macrophages and their coreceptor/ligands) and how their signaling state in disease relates to clinical outcomes.

IV. To store and/or analyze surplus blood or tissue including bone marrow, if available, for potential future exploratory research into factors that may influence development of AML and/or response to the combination (where response is defined broadly to include efficacy, tolerability or safety).

OUTLINE: This is a phase Ib, dose-escalation study of venetoclax and magrolimab followed by a phase II study.

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) over 30-60 minutes on days 1-7, venetoclax orally (PO) once daily (QD) on days 1-28 of cycle 1 (may be reduced to days 1-21 for subsequent cycles after principal investigator approval), and magrolimab IV over 2-3 hours on days 1, 4, 8, 11, 15, and 22 of cycle 1, days 1, 8, 15, and 22 of cycle 2, and days 1 and 15 of cycle 3 and subsequent cycles. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1) WHO diagnosis of AML (excluding acute promyelocytic leukemia (APL)
* Phase Ib dose finding cohort: Participants aged ≥18 years old with relapsed/refractory AML are eligible if they are not eligible for potentially curative therapy such as effective salvage therapy or hematopoietic stem cell transplantation or who refuse these options at the time of enrollment. Participants must have received at least one prior therapy for AML. Participants may have received up to 2 prior therapies for AML (i.e. up to salvage 2 status allowed). Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2
* Phase II (frontline cohort): Participants with newly diagnosed AML who are chemonaive (specified in 4.1.5) who are ineligible for intensive chemotherapy based on EITHER:

A. ≥75 years of age OR

B. <75 years of age with at least 1 of the following relevant comorbidities:

* Poor performance status (ECOG) score of 2.
* Clinically significant heart or lung comorbidities, as reflected by at least 1 of:

  1. Left ventricular ejection fraction (LVEF) ≤50%.
  2. Lung diffusing capacity for carbon monoxide (DLCO) ≤65% of expected.
  3. Forced expiratory volume in 1 second (FEV1) ≤65% of expected.
  4. Chronic stable angina or congestive heart failure controlled with medication.
  5. Creatinine clearance ≥ 30 mL/min to < 45 ml/min calculated by the Cockcroft-Gault formula or measured by 24 hours' urine collection
* Other contraindication(s) to anthracycline therapy (must be documented).
* Other comorbidity the investigator judges incompatible with intensive remission induction chemotherapy, which must be documented and approved by the PI."

For participants with prior MDS or chronic myelomonocytic leukemia (CMML) or MPN who transformed to AML, therapy received for MDS, CMML, or MPN is NOT considered as prior therapy for AML. Participants with MDS or CMML treated with HMA therapies who progress to AML, and have no available therapies or are not candidates for available therapies, will be eligible to be enrolled to the relapsed/refractory cohort at the time of progression to AML. Temporary prior measures such as apheresis, ATRA, steroids while diagnostic work-up of AML is being performed are allowed and not counted as a prior salvage

* Phase II (relapsed/refractory prior venetoclax naïve cohort): Participants aged ≥18 years old with relapsed/refractory AML are eligible if they are not eligible for potentially curative therapy such as effective salvage therapy or hematopoietic stem cell transplantation or who refuse these options at the time of enrollment. Participants must have received at least one prior therapy for AML or at least one prior HMA therapy for MDS/CMML or MPN. Participants may have received up to 2 prior therapies for AML (i.e. up to salvage 2 status allowed). Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2. Participants must not have received prior venetoclax for MDS or AML.
* Phase II (relapsed/refractory prior venetoclax exposed cohort): Participants aged ≥18 years old with relapsed/refractory AML are eligible if they are not eligible for potentially curative therapy such as effective salvage therapy, targeted therapies, or hematopoietic stem cell transplantation or who refuse these options at the time of enrollment. Participants must have received at least one prior therapy for AML or at least one prior HMA therapy for MDS/CMML or MPN. Participants may have received up to 1 prior therapies for AML (i.e. up to salvage 1 status allowed). Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2. Participants must have received prior venetoclax for MDS or AML.

  * Participants with newly diagnosed AML with poor risk karyotype or complex karyotype per ELN2017 and/or TP53 deletions/mutations of any age >/=18 years of age will be eligible for the Phase II (frontline cohort) regardless of eligibility or fitness for intensive chemotherapy
  * For Phase II (frontline cohort): Participants must be chemonaïve, i.e., not have received any chemotherapy (except hydrea or up to 2 doses of ara-C for transient control of hyperleukocytosis) for AML. They may have received transfusions, hematopoietic growth factors or vitamins for an antecedent hematological disorder (AHD) or for AML. Temporary prior measures such as apheresis, ATRA, steroids or hydrea while diagnostic work-up is being performed are allowed and not counted as a prior salvage. Supportive care therapy for MDS (growth factors, transfusions) will not be considered as prior therapy for MDS/AML and these participants will be enrolled to the frontline cohort of the study if they are otherwise eligible.
  * In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of protocol therapy will be at least 2 weeks or at least 5 half-lives (whichever is shorter). The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochure's, or drug-administration manuals) and will be documented in the protocol eligibility document. The toxicity from prior therapy should have resolved to Grade ≤1, however alopecia and sensory neuropathy Grade ≤2 not constituting a safety risk based on investigators judgement is acceptable. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions: (1) intrathecal (IT) therapy for patients with controlled CNS leukemia at the discretion of the PI. (2) Use of up to 2 doses of cytarabine (up to 2 g/m2 each dose) for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy. Since the effect of most IO-agents, HMA-therapies, venetoclax may be delayed, use of hydroxyurea for patients with rapidly proliferative disease is allowed on study and before the start of study therapy and will not require a washout. These medications will be recorded in the case-report form.
  * Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS disease is permitted. Participants with a known history of CNS disease or leukemic brain metastasis must have been treated locally, have at least 2 consecutive LPs with no evidence of CNS leukemia at the time of enrollment, and must be clinically stable for at least 4 weeks prior to enrollment and have no ongoing neurological symptoms that in the opinion of the treating physician are related to the CNS disease (sequelae that are a consequence of the treatment of the CNS disease are acceptable).
  * Serum biochemical values with the following limits:

Participants must have adequate renal function as demonstrated by a creatinine clearance (CrCl) ≥ 30 mL/min calculated by the Cockcroft-Gault formula or measured by 24 hours' urine collection.

For participants with BMI >23, Adjusted body weight and not Ideal Body Weight is the recommended parameter (Winter et al, Pharmacotherapy. 2012 Jul; 32(7):604-12; Brown et al, Ann Pharmacother. 2013 Jul-Aug;47(7-8): 1039-44).

* Total bilirubin <1.5 x ULN unless considered due to Gilbert's syndrome,
* Aspartate aminotransferase or alanine aminotransferase ≤2.0 x ULN (aspartate aminotransferase or alanine aminotransferase ≤3.0 x ULN if deemed related to leukemia by the treating physician)
* White blood cell count <15 x 109/L. Participants must have a WBC count <15 x 109/L prior to each dose of magrolimab in Cycle 1. Hydroxyurea may be used to reduce the WBC count to ≤15x109/L.
* Ability to understand and provide signed informed consent.
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment.
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 4 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment.

Adequate methods of contraception include:

* Total abstinence when this is in line with the preferred and usual lifestyle of the participants. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participants
* Combination of any of the two following (a+b or a+c or b+c)

  1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository In case of use of oral contraception, women should have been stable on the same pill before taking study treatment.

Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction.

Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

Male participants who are sexually active with a WOCBP and who have not had vasectomies must be willing to use a barrier method of contraception during the study and for 3 months after the last dose of magrolimab, venetoclax or azacitidine, whichever ends later.

Women who are pregnant or breastfeeding will not be eligible.

Exclusion Criteria:

* Participants with known allergy or hypersensitivity to magrolimab, venetoclax, azacitidine or any of their components.
* Participants with any other known concurrent severe and/or uncontrolled medical condition including but not limited to diabetes, cardiovascular disease including hypertension, renal disease, or active uncontrolled infection, which could compromise participation in the study. Participants on active antineoplastic or radiation therapy for a concurrent malignancy at the time of screening. Maintenance therapy, hormonal therapy, or steroid therapy for well-controlled malignancy is allowed.
* Prior organ transplantation including allogenic stem-cell transplantation within 3 months prior to planned enrollment, active graft versus host disease (GVHD) >Grade 1, or requiring transplant-related immunosuppression, excluding prednisone 10mg or equivalent steroid.
* Known inherited or acquired bleeding disorders
* Prior treatment with a CD47 or SIRP targeting agent.
* Participants with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia.
* Participants with a known HIV infection that is not well controlled (i.e. any detectable circulating viral load) at the time of enrollment.
* Participants with known positive hepatitis B or C infection by serology, with the exception of those with an undetectable viral load within 3 months (Hepatitis B or C testing is not required prior to study entry). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+] may participate.
* Patients who have consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
* Participants who have had any major surgical procedure within 14 days of Day 1.
* Other severe acute or chronic medical conditions that is active and not well controlled including colitis, inflammatory bowel disease, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Active and uncontrolled disease (active infection requiring systemic therapy or fever likely secondary to infection within prior 48 hours): prophylactic antibiotics or prolonged course of IV antibiotics for controlled infection are allowed, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure NYHA class III/IV, clinically significant and uncontrolled arrhythmia) as judged by the treating physician.
* Participants unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of the combination drugs (phase Ib) | 28 days
Response rate (complete remission + complete remission with incomplete count recovery) (phase II) | Within 3 months of treatment initiation
  Will be monitored simultaneously. Will be estimated along with 95% credible intervals. Chi-square tests or Fisher's exact test will be used to evaluate the association between patient's prognostic factor and response.
Incidence of adverse events (phase II) | Within 3 months of treatment initiation
  Toxicities are defined as drug-related non-hematological grade >= 3 adverse events.
Event-free survival (phase II) | Time duration from the start of treatment to disease progression/death or censored at last follow-up while on the drug, assessed up to 100 days
  Kaplan-Meier method will be used.
Duration of response (phase II) | Up to 100 days
  Kaplan-Meier method will be used.
Overall survival (phase II) | Up to 100 days
  Kaplan-Meier method will be used.

SECONDARY OUTCOMES:
Change in gene expression (phase II) | Baseline up to 100 days
  Paired t-tests will be used.
Change in clinical variables (phase II) | Baseline up to 100 days
  Paired t-tests will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Naval G Daver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04435691/ICF_000.pdf